CLINICAL TRIAL: NCT04111549
Title: Rehabilitation of Executive Function in Aging Veterans With History of TBI
Brief Title: GOALS Cognitive Training Delivered to Aging Veterans in Person or Via Telehealth
Acronym: TeleGOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E3073-W; 1IK2RX003073-01A2 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Brain Injuries, Traumatic; Executive Dysfunction
Keywords: Veterans; Rehabilitation; Cognitive training; Telehealth
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: After a 5-week delay repeat baseline, participants will be randomized to receive either in-person GOALS or GOALS delivered via home-based video telehealth.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to which condition (in-person or home-based telehealth) a participant completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based telehealth GOALS (Experimental): Participants in this arm will receive the GOALS intervention via in-home video telehealth.
  Interventions: Other: Home-based telehealth GOALS
- In-person GOALS (Active Comparator): Participants in this arm will receive the GOALS intervention in the traditional in-person format.
  Interventions: Other: In-person GOALS

INTERVENTIONS:
Other: Home-based telehealth GOALS — Goal Oriented Attentional Self-Regulation (GOALS) is a manualized cognitive training intervention for problems with attention and executive control that has been shown to improve cognitive, emotional, and functional outcomes in civilians and Veterans with history of TBI, including Veterans 65 and older, and healthy older adults. It will be delivered to aging Veterans with history of TBI via in-home video telehealth.
  Arms: Home-based telehealth GOALS
Other: In-person GOALS — Goal Oriented Attentional Self-Regulation (GOALS) is a manualized cognitive training intervention for problems with attention and executive control that has been shown to improve cognitive, emotional, and functional outcomes in civilians and Veterans with history of TBI, including Veterans 65 and older, and healthy older adults. It will be delivered to aging Veterans with history of TBI in person.
  Arms: In-person GOALS

SUMMARY:
This study will use technology to deliver effective treatment for cognitive problems associated with TBI to Veterans at home, which may result in improved daily functioning and increased access to health care for the growing population of aging Veterans with history of TBI. The successful completion of this project may also increase older Veterans' ability to participate in research through increased understanding of the effect of in-home research opportunities on recruitment and retention. Additionally, the evidence gathered from this study may be used in future research studying home-based cognitive rehabilitation treatments for Veterans using telehealth technology.

DETAILED DESCRIPTION:
The goal of this project is to investigate the feasibility and acceptability of using technology to implement home-based executive function training for aging Veterans with history of traumatic brain injury (TBI).

Background: Problems with attention and executive control are some of the most common sequelae of TBI, and these areas of cognition are also known to be vulnerable to aging. Goal Oriented Attentional Self-Regulation (GOALS) is a manualized cognitive training intervention for problems with attention and executive control that has been shown to improve cognitive, emotional, and functional outcomes in civilians and Veterans with history of TBI, including Veterans 65 and older, and healthy older adults.

Relevance and significance to Veteran's health: TBI is prevalent among Veterans. Home-based telehealth (HBT) may be an effective tool to address lack of access to health care for aging Veterans.

Aim 1: Complete adaptation of the IP-GOALS protocol for a) HBT use and b) use with older Veterans via collection of feedback from [n=8] Veterans 65+ with history of TBI and cognitive complaints. Aim 2: Examine the feasibility (defined as recruitment yield, dropout after randomization, retention, and adherence) and participant-rated acceptability of [IP and] HBT-GOALS in n=36 Veterans 65+ with history of TBI and cognitive complaints. Hypothesis 2: Feasibility will be demonstrated by achieving targeted recruitment goals with reasonable rates of dropout after randomization, retention, and adherence, and high levels of participant-rated acceptability in both groups. Aim 3: Estimate effect sizes for [HBT-GOALS and IP-GOALS using a double-baseline control] on improving a) cognitive performance and self-reported b) emotional regulation and c) daily functioning in the same Aim 2 study cohort to inform sample size requirements for a future clinical trial. Hypothesis 3: Effect size estimates will provide evidence of clinically meaningful improvement on a) cognitive functioning (Attention and Executive Function Composite), b) emotional regulation (Profile of Mood States Total Mood Disturbance Score), and c) daily functioning outcomes (Mayo-Portland Adaptability Inventory Total Score). Exploratory analysis a) will examine whether Veteran characteristics (e.g., age, sex, family/caregiver support, distance to nearest clinic, and health/mobility issues including chronic pain) are associated with differences in participant-rated acceptability and feasibility (i.e., recruitment yield, dropout after randomization, retention and adherence), and [response to IP/HBT-GOALS vs. double baseline control.] Exploratory analysis b) will examine distribution of responses to select criteria to define responders in future studies.

Methods: Adaptation phase (Aim 1): Adaptation of the existing GOALS protocol for a) HBT use and b) use with older Veterans will be completed by collecting post-training feasibility and acceptability data. Pilot phase (Aims 2 and 3 and Exploratory Analyses): Feasibility, acceptability, cognitive, emotional, and daily functioning data will be collected from n=36 Veterans 65 or older before (baseline and delay baseline) and after participation in GOALS training delivered in person (IP) or via HBT. Veterans will be randomly assigned to IP or HBT. Outcome measures include participant-rated acceptability; feasibility (i.e., recruitment yield, dropout after randomization, retention, and adherence); standardized and validated measures of neurocognitive functioning; self-report of symptoms of depression, PTSD, mood disturbance, and daily functioning.

Innovation: The proposed study is the first to investigate implementation of an established cognitive rehabilitation intervention for use with aging Veterans with history of TBI and delivery via in-home videoconferencing technology.

Implications: This research may promote improved daily functioning for aging Veterans with history of TBI through rehabilitation of executive function, and increase access to such treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 65 or older with history of chronic TBI (>6 months post-injury) -- sustained either during military service

  * including in combat
  * or as a civilian
* Self-reported cognitive complaints [1 moderate or severe cognitive symptom(s) on the Neurobehavioral Symptom Inventory (NSI [58]) that interfere(s) with daily function]
* Endorsement of comfort and familiarity with technology and/or the possession of a personal computer, or other HBT-compatible device

  * i.e., tablet, or smartphone
* Per the investigators' preliminary patient survey, approximately 75% of the target population has access to a personal computer

  * Participants who do not endorse comfort/familiarity with technology may be eligible to participate if they can identify a family member or other caregiver who is consistently present and willing to assist with connecting to study sessions
* A limited number of VA-issued tablets will be available for use by participants who do not have access to a personal computer or other HBT-compatible device

Exclusion Criteria:

Moderate-severe objective cognitive impairment, as measured by score <20 on the Montreal Cognitive Assessment (MoCA [59-61]), that interferes with daily functioning (i.e., Major Neurocognitive Disorder)

* Unstable medical, neurologic, or psychiatric conditions precluding participation in research activities
* Other reasons for being unable or unwilling to participate in study procedures
* Ongoing illicit or prescription drug (Mini International Neuropsychiatric Interview Version 7.0.2 (MINI) [79] or alcohol abuse (Alcohol Use Disorders Test-Consumption (AUDIT-C) [62]>8)
* Active psychosis
* Poor English comprehension

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Attention and Executive Function Change | Baseline, after 5 week delay repeat baseline, and after 5 week intervention
  Composite of neuropsychological measures of attention and executive function: Letter Number Sequencing; Auditory Consonant Trigrams 9, 18, 36 sec; Digit Vigilance Test -Time & Errors; Trails B; DKEFS Stroop Inhibition Time & Errors; DKEFS Stroop Inhibition-Switching Time & Errors; DKEFS Verbal Fluency Switching; & DKEFS Design Fluency Switching. All scores will be transformed to z scores using published normative data and then an average will be calculated to obtain the single Overall Attention and Executive Function score. The composite z score will range from -3 to 3, with higher scores indicating better performance.
Profile of Mood States (POMS) Total Mood Disturbance Change | Baseline, after 5 week delay repeat baseline, and after 5 week intervention
  Measure of emotion regulation and overall psychological distress. Scores range from 0-200, and higher scores indicate more distress.
Mayo-Portland Adaptability Inventory Total Score Change | Baseline, after 5 week delay repeat baseline, and after 5 week intervention
  Post-TBI daily functioning: abilities and participation in daily activities. Scores range from 0-111, with lower scores indicating better function and greater ability and participation.

CONTACTS AND LOCATIONS:
Overall Officials: Erica S. Kornblith, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04111549/ICF_000.pdf